CLINICAL TRIAL: NCT01044927
Title: Phase 3 Clinical Trial Studying the Efficacy of a Proactive Integrated Approach to Care in Patients With Advanced COPD
Brief Title: Advanced eHealth for Chronic Obstructive Pulmonary Disease (COPD) in Colorado
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Department of Public Health and Environment (Other Government); Kaiser Permanente (Other); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-0587; 07 FLA 00834 (Other: CDPHE)
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; telemedicine; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Delivery of Health Care, Integrated; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proactive Integrated Care (Experimental): COPD-specific education, self-management instruction, remote monitoring and enhanced communication with a coordinator
  Interventions: Other: Integrated Care
- Standard Care Control (Active Comparator): No intervention other that measurements taken at 0, 3, 6 and 9 months of the study.
  Interventions: Other: Standard Therapy

INTERVENTIONS:
Other: Integrated Care — Comparison of the effect of COPD education, self-management instruction, home monitoring with a Health Buddy Telemonitor, pulse oximeter, pedometer and spirometer, and enhanced communication with a study coordinator (cell phone access)
  Arms: Proactive Integrated Care
Other: Standard Therapy — No intervention was made. Data measurements were taken at 0, 3, 6 and 9 months, as in the active intervention group.
  Arms: Standard Care Control

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is the 4th leading cause of death in the United States, affects 24 million people and is responsible for up to $32 billion annually in direct and indirect health care costs. Based upon these national COPD prevalence data, we estimate that 483,000 Coloradans have COPD (193,000 diagnosed and 290,000 undiagnosed), and that the care of these patients costs up to $490 million annually. Therefore, to alter the impact of COPD on the State and People of Colorado, we propose to introduce a telephone-dependent, internet-supported, self-monitoring "eHealth" management system in both urban and rural Colorado settings in order to decrease healthcare utilization, improve the management of COPD based upon current national guidelines, improve quality of life, reduce health care costs decrease COPD exacerbations. We base this program on a successful clinical pilot study, performed at the University of Colorado Hospital (UCH) during 2004-2005, which demonstrated dramatic improvements in quality of life and decreased health care costs. We propose to enroll patients with advanced COPD, or a history of COPD exacerbations, because these are the patients with the highest healthcare costs, the greatest disability, and the highest mortality. The ultimate goal of this project is to demonstrate the feasibility and efficacy of this proactive management strategy as it is disseminated throughout urban and rural Colorado. In this first phase we will target two Denver Metro sites, UCH and Kaiser-Permanente (KP), and rural sites (to be determined). We chose these urban sites because of their strong interest in enacting the eHealth Program, because of their organized systems of healthcare delivery and because of the numbers of COPD patients that they serve. We are particularly enthusiastic about the application of this technology to rural, underserved areas, because this approach has the potential to dramatically improve delivery of healthcare to a large portion of Colorado that is chronically plagued by inadequate health care networks and lack of specialty care. More broadly, we are enthusiastic about the prospect that eHealth programs may hold the potential to improve healthcare delivery for many chronic illnesses, in addition to COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD Diagnosis per GOLD Guidelines
* Airflow obstruction on spirometry defined as an FEV1/FVC less than or equal to 70% and an FEV1 less than or equal to 50% predicted, or an FEV1 greater than 50% predicted with a history of a COPD exacerbation within the previous year.
* Standard telephone access
* US Citizen and Colorado resident

Exclusion Criteria:

* Asthma
* Co-existing conditions that are likely to cause death within two years, CXR evidence of interstitial lung disease or other pulmonary diagnoses at the time of enrollment, end-stage liver disease, end-stage renal disease, end-stage muscle disease, HIV disease or dementia.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2006-09; Primary Completion 2007-08 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Healthcare utilization | 9 months

SECONDARY OUTCOMES:
Quality of Life by St. Georges Respiratory Questionnaire | 3, 6 and 9 months
Guideline-based medical therapy | 9 months
Exercise capacity | 9 months
Oxygen utilization and pre-and post-exercise oxygen saturations | 9 months
Body Mass Index, Obstruction, Dyspnoea, Exercise Capacity (BODE) index | 9 months
Symptoms including cough, sputum production and dyspnea (modified Medical Research Council (MMRC) MMRC Dyspnea Scale) | 9 months
Smoking status | 9 months
Pulmonary rehabilitation | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: William Vandivier, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Kaiser Permanente, Denver, Colorado